CLINICAL TRIAL: NCT06967805
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of MTX-463 in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: WISPer: Evaluation of MTX-463 in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mediar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTX-463-I201; 2025-521278-32 (EudraCT Number); WISPer (Other: Mediar Therapeutics)
Record Dates: First submitted 2025-04-14; First posted 2025-05-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: MTX-463-I201; MTX-463; IPF; Idiopathic Pulmonary Fibrosis; Adult; Fibrosis; Monoclonal Antibody; MAB; FVC; WISPer
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MTX-463 (Experimental): MTX-463
  Interventions: Biological: MTX-463
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MTX-463 — MTX-463 is an immunoglobin G1 (IgG1) monoclonal antibody directed against WNT-inducible signaling pathway protein 1 (WISP1). WISP1 (aka CCN-4) is a matricellular protein that appears to be upregulated locally in response to certain chronic diseases, including IPF, and malignancies.
  Arms: MTX-463
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Phase 2a, Randomized, Double-blind, Placebo-Controlled Study of the Safety and Efficacy of MTX-463 in Participants with Idiopathic Pulmonary Fibrosis (IPF)

DETAILED DESCRIPTION:
Participants with IPF who meet the study's inclusion and exclusion criteria will be randomly assigned in a 1:1 ratio to receive MTX-463 or a matching placebo by intravenous (IV) infusion. Concomitant use of one of the approved IPF therapies, pifenidone or nintedanib, is permitted, and it is expected that about half the study population will be on one of those medications. Participants randomized to the MTX-463 arm of the study will receive an IV infusion every 4 weeks, beginning at Day 0 and ending at Week 20. The End of Treatment Visit will occur at Week 24, 4 weeks after the final infusion; and a final Safety Follow-Up Visit will occur at Week 28, 8 weeks after the final infusion. Assessments of FVC will occur at Screening, Baseline, and at all subsequent treatment visits up to and including Week 24. L-PF assessments will be performed at Baseline and Week 24. Participants will have blood drawn for safety assessment and to assess WISP1 levels at Baseline and every 4 weeks throughout the study. Blood will be drawn for serum PK analyses relative to the first and last doses of MTX-463.

ELIGIBILITY:
Inclusion Criteria:

* Participants with IPF of any gender ≥ 40 years of age at time of signing the informed consent.
* Able to understand the study and provide signed, written informed consent.
* Able to read and understand the language of the informed consent and other trial-related materials.
* Meet the American Thoracic Society, European Respiratory Society, Japanese Respiratory Society, and Latin American Thoracic Association (ATS/ERS/JRS/ALAT) 2019 criteria for the diagnosis of IPF; Diagnosed with IPF within 7 years of screening.
* If a participant is on treatment with pirfenidone or nintedanib, the dose of the medication must be stable for ≥ 90 days prior to Screening with plans to maintain the same dose throughout the study treatment period. Use of both agents together is not permitted.
* If a participant was on treatment with nintedanib or pirfenidone, and the agent has been discontinued, this must have occurred ≥ 30 days prior to Screening. At Screening, there must also be no plan to start either of these medications for the duration of the study.
* FVC of ≥ 45 percent predicted (pp) at screening.
* DLCO of ≥ 25pp at screening.
* Willing and able to complete all protocol required study visits and procedures.
* All participants of childbearing potential must have a negative serum pregnancy test at Screening.
* Participants with reproductive potential must agree to use and follow medically approved contraceptive precautions during the study

Exclusion Criteria:

* Acute exacerbation of IPF within 6 months of Screening or during the Screening Period.
* Forced expiratory volume in 1 second (FEV1)/FVC ratio of <0.7 at Screening.
* Requirement for continuous supplemental oxygen. Intermittent supplemental oxygen use (e.g., during exercise or sleep) is permitted.
* Expected to receive a lung transplant within the study duration.
* Current active bacterial infection or use of antibiotics for suspected lung infection in the 30 days prior to Screening.
* Planned surgery within the study duration.
* Clinically significant pulmonary hypertension.
* Use of immunosuppressive therapy (excluding corticosteroids). If previously on such agents, they should have been discontinued for at least 5 half-lives or 90 days, whichever is longer, prior to Screening.
* Use of systemic corticosteroids (prednisone or equivalent) at a dose ≥ 10 mg once daily within 30 days of Screening.
* Currently smoking or vaping.
* Current known malignancy, or history of cancer, or lymphoproliferative disorder other than non-melanomatous skin cancers, within 2 years of Screening.
* Current infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Currently pregnant, breast feeding, or planning to conceive for the length of the study.
* History of severe depression, psychosis, or suicidal ideation, as determined by the Investigator, within 2 years of Screening.
* Any clinically significant disease or laboratory abnormality detected at Screening that might interfere with a participant's ability to complete the study, on-study evaluations, or participant safety.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2× upper limit of normal (ULN) at Screening.
* Any other concurrent active medical condition determined by the Investigator to interfere with participant's ability to complete the trial.
* Known allergy to MTX-463 or any of its excipients.
* Any prior use of MTX-463 or other therapy targeting WISP1.
* Any other concurrent experimental agent or an active part of any other clinical trial, unless they have stopped taking the investigational product at least 5 half-lives or 30 days before Screening, whichever is longer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of MTX-463 on the change from Baseline in forced vital capacity (FVC) | 24 Weeks
  Change from Baseline to Week 24 in Forced Vital Capacity (FVC)

SECONDARY OUTCOMES:
To assess the safety and tolerability of MTX-463 in participants with IPF, as measured by incidence of treatment emergent adverse events | 28 Weeks
  Incidence of treatment-emergent adverse events (TEAEs) from Baseline until Week 28 in each group
To assess the safety and tolerability of MTX-463 in participants with IPF, as measured by incidence of treatment related adverse events | 28 Weeks
  Incidence of treatment related adverse events from baseline until Week 28 in each group
To assess the safety and tolerability of MTX-463 in participants with IPF, as measured by incidence of serious treatment emergent adverse events | 28 Weeks
  Incidence of serious treatment emergent adverse events from baseline until Week 28 in each group
To assess the safety and tolerability of MTX-463 in participants with IPF, as measured by incidence of severe treatment emergent adverse events | 28 Weeks
  Incidence of severe treatment emergent adverse events from Baseline until week 28 in each group
To assess the safety and tolerability of MTX-463 in participants with IPF, as measured by incidence of treatment emergent abnormalities on clinical laboratory tests | 28 Weeks
  Incidence of treatment emergent abnormalities on clinical laboratory tests from baseline until Week 28 in each group
To assess the safety and tolerability of MTX-463 in participants with IPF, as measured by incidence of abnormal findings on physical exam | 28 Weeks
  Incidence of abnormal findings on physical exam from baseline until Week 28 in each group
To assess the safety and tolerability of MTX-463 in participants with IPF, as measured by incidence of treatment discontinuations | 28 Weeks
  Incidence of treatment discontinuations from baseline until Week 28 in each group
To assess the effect of MTX-463 on the change from Baseline in the percent predicted FCV (FVCpp) | 24 Weeks
  Change from Baseline to Week 24 in the percent predicted FVC (FVCpp)
To collect sparse pharmacokinetics (PK) of MTX-463 in participants with IPF | 24 Weeks
  Samples will be collected from baseline until Week 24 to assess the trough serum concentrations of the study drug

OTHER OUTCOMES:
To assess the development of antidrug antibodies (ADA) against MTX-463 | 28 Weeks
  Samples will be collected from baseline until Week 28 to assess the rate at which antibodies develop to the study drug
To assess the effect of MTX-463 on the change from Baseline in FVC in participants on concomitant nintedanib or pirfenidone | 24 Weeks
  The change from baseline to week 24 in the mean FVC (in ML) will be measured in each group in the subset of participants who enter the study on background IPF medications, pirfenidone or nintedanib
To assess the effect of MTX-463 on the change from Baseline in FVC in participants not on concomitant nintedanib or pirfenidone | 24 Weeks
  The change from baseline to week 24 in the mean FVC (in ML) will be measured in each group in the subset of participants who enter the study not on any background IPF medications, pirfenidone or nintedanib
To assess the effect of MTX-463 on the change from Baseline in the Living with Pulmonary Fibrosis (L-PF) Questionnaire total score | 24 Weeks
  Change from Baseline to Week 24 in L-PF total score. The L-PF is scored on a scale of 0-100, with higher numbers indicating greater impairment.
To assess whether serum WNT-inducible signaling pathway protein 1 (WISP1) levels at Screening predict improved outcomes with MTX-463 treatment | 24 Weeks
  * Change from Baseline to Week 24 in total WISP1 levels
  * Change from Baseline to Week 24 in free WISP1 levels
  * Change from Baseline to Week 24 in FVC by free and total WISP1 screening quartiles
To assess the effect of MTX-463 on the change from Baseline in percent predicted diffusing capacity of the lungs for carbon monoxide (DLCO) | 24 Weeks
  Change from Baseline to Week 24 in percent predicted DLCO
To evaluate the time to disease progression as determined by change in FVC, IPF-related changes, or death | 28 Weeks
  Time to disease progression with progression being defined as ≥10% decline in FVC from Baseline, IPF related hospitalization, or death
To assess the effect of MTX-463 on Pro-C3 | 24 Weeks
  The mean change from baseline to week 24 in the level of ProC3, a biomarker of IPF, in the serum will be measured in each group
To assess the effect of MTX-463 on interleukin-6 | 24 Weeks
  The mean change from baseline to week 24 in the level of interleukin-6 (IL-6), a biomarker of IP, in the serum will be measured in each group

CONTACTS AND LOCATIONS:
Overall Officials: Todd Astor, MD, Study Chair — Mediar Therapeutics
Locations (44):
- United States (22):
  - WISPer Site in Birmingham, AL, Birmingham, Alabama
  - WISPer site in Phoenix, AZ, Phoenix, Arizona
  - WISPer Site in Los Angeles, CA, Los Angeles, California
  - WISPer site in Newport Beach, CA, Newport Beach, California
  - WISPer Site in Palm Springs, CA, Palm Springs, California
  - WISPer Site in Denver, CO, Denver, Colorado
  - WISPer site in Loxahatchee, FL, Loxahatchee Groves, Florida
  - WISPer site in Champaign, IL, Champaign, Illinois
  - WISPer site in Kansas City, KS, Kansas City, Kansas
  - WISPer site in Shreveport, LA, Shreveport, Louisiana
  - WISPer Site in Baltimore, MD, Baltimore, Maryland
  - WISPer Site in Ann Arbor, MI, Ann Arbor, Michigan
  - WISPer Site in Detroit, MI, Detroit, Michigan
  - WISPer site in New York, NY, New York, New York
  - WISPer Site in Durham, NC, Durham, North Carolina
  - WISPer site in Greensboro, NC, Greensboro, North Carolina
  - WISPer site in Oklahoma City, OK, Oklahoma City, Oklahoma
  - WISPer Site in Charleston, SC, Charleston, South Carolina
  - WISPer Site in Nashville, TN, Nashville, Tennessee
  - WISPer site in Dallas, TX, Dallas, Texas
  - WISPer Site in Salt Lake City, UT, Salt Lake City, Utah
  - WISPer Site in Wilwaukee, WI, Milwaukee, Wisconsin
- Australia (4):
  - WISPer site in Greenslopes, Australia, Greenslopes
  - WISPer site in Melbourne, Australia, Melbourne
  - WISPer site in Midland, Australia, Midland
  - WISPer site in Westmead, Australia, Westmead
- WISPer Site in Brussels, Belgium, Brussels, Belgium
- WISPer Site in Belo Horizonte, Brazil, Belo Horizonte, Brazil
- Canada (3):
  - WISPer Site in Calgary, Alberta, Calgary, Alberta
  - WISPer site in Ajax, ON, Ajax, Ontario
  - WISPer site in Trois-Rivières, Quebec, Trois-Rivières, Quebec
- WISPer Site in Split, Split, Croatia
- France (3):
  - WISPer Site in Nice, France, Nice
  - WISPer Site in Paris, France, Paris
  - WISPer Site in Rennes, France, Rennes
- Ireland (3):
  - WISPer Site in Drogheda, Ireland, Drogheda
  - WISPer Site in Dublin, Ireland, Dublin
  - WISPer Site in Letterkenny, Ireland, Letterkenny
- Spain (2):
  - WISPer Site in Barcelona, Spain, Barcelona
  - WISPer Site in Madrid, Spain, Madrid
- United Kingdom (4):
  - WISPer Site in Birmingham, UK, Birmingham
  - WISPer Site in Cambridge, UK, Cambridge
  - WISPer Site in Edinburgh, UK, Edinburgh
  - WISPer Site in Oxford, UK, Oxford

IPD SHARING:
Plan to Share IPD: No